CLINICAL TRIAL: NCT02821897
Title: Value of Target-controlled Intravenous Anaesthesia (TCIVA) to Optimize Coverage of the Low Back Pain Territory in Patients With Chronic Refractory Postoperative Multifocal Low Back and Legpain
Brief Title: Value of Target-controlled Intravenous Anaesthesia (TCIVA) in Spinal Cord Stimulation
Acronym: AIVOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIVOC
Record Dates: First submitted 2016-06-27; First posted 2016-07-04 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Target-controlled Intravenous Anaesthesia (Experimental): Patients have a target controlled intravenous anaesthesia to implant the spinal cord stimulation lead with active cooperation during the surgery.
  Interventions: Procedure: Target-controlled intravenous anaesthesia
- Total anesthesia (Active Comparator): Patients have a total anaesthesia to implant the spinal cord stimulation lead without active cooperation during the surgery.
  Interventions: Procedure: Total anaesthesia

INTERVENTIONS:
Procedure: Target-controlled intravenous anaesthesia
  Arms: Target-controlled Intravenous Anaesthesia
Procedure: Total anaesthesia
  Arms: Total anesthesia

SUMMARY:
Study design 60 patients Monocenter prospective study Randomized in 2 groups 36 months Objectives Demonstrate the superiority of target controlled intravenous anesthesia versus total anesthesia with the low back paresthesia mapping in at least 95% of patients implanted with a multicolumn lead.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and ≤ 80 years
* FBSS
* Radicular leg et lumbar pain
* For more than 3 months after one or many spine surgeries
* Mixt pain (radicular leg et lumbar) with Neuropathic status
* Failure of conservative treatment
* Severe uni or bilateral radicular pain > 5 / 10

Exclusion Criteria:

* Age <18 years and> 80 years.
* BMI > 30 kg/m2.
* Back pain that can be treated by surgery (discogenic, vertebral instability, …)
* Contraindication to TCIVA anesthesia under propofol remifentanil
* Psychiatric status
* Cancer
* No signature of informed consent.
* Women of childbearing without contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Postoperative paresthesia coverage >= 50% of the lower lumbar determined using a paresthesia cover mapping | 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, Worldwide, France